CLINICAL TRIAL: NCT07053540
Title: Investigation of the Impact of Video Games and Various Activities on the Success of Videolaryngoscopy
Brief Title: Impact of Video Games and Activities on Videolaryngoscopy Success
Status: Enrolling by invitation | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ali Genc, Assistant professor, Tokat Gaziosmanpasa University
Other Study IDs: 25-MOBAEK-214
Record Dates: First submitted 2025-06-19; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: The Effects of Video Game Playing Habits and Some Sports Activities on Intubation Performance With Video Laryngoscopy
Keywords: Intubation; videolaryngoscopy; video games

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Those who regularly play video games or do some sports activities: Video games and certain athletic activities are tasks that require active hand-eye coordination and the ability to think three-dimensionally. It is suggested that activities such as videolaryngoscopy, which depend on hand-eye coordination, motor skills, visual attention, and spatial awareness, may be influenced by experiences gained through video gaming and similar activities.
- Those who do not play video games or do certain sports activities: Activities such as playing video games or engaging in certain sports that require hand-eye coordination and three-dimensional thinking are not regularly performed by some individuals. It is hypothesized that activities involving hand-eye coordination, motor skills, visual attention, and spatial awareness-such as video gaming or specific physical activities-may positively influence these skills in tasks like videolaryngoscopy and other procedures demanding similar competencies.

SUMMARY:
This study aims to investigate the factors influencing the videolaryngoscopy success among fourth-year medical students participating in anesthesia clerkship. Specifically, it examines the impact of activities such as video gaming and various other hobbies on fundamental skills related to videolaryngoscopy, including hand-eye coordination, motor skills, visual attention, and spatial awareness. In this context, the study evaluates how regular engagement in activities such as video games, sports, chess, Rubik's Cube, 3D puzzles, arts and crafts, and playing musical instruments may contribute to intubation success, intubation duration, and the quality of glottic visualization.

DETAILED DESCRIPTION:
Research will include fourth-year students who are volunteering and have no prior endotracheal intubation experience, during the 2025-2026 academic year at Tokat Gaziosmanpaşa University Faculty of Medicine's Department of Anesthesiology. Students with previous clinical airway management experience-such as videolaryngoscopy (VL) or direct laryngoscopy intubation-will be excluded, particularly those unable to utilize VL due to motor impairments (e.g., neuromuscular disorders) or recent hand surgeries. Students will be enrolled after receiving information about the study and providing informed consent.

Prior to participation, all students will receive theoretical training on airway management and videolaryngoscopy-assisted intubation. Following the theoretical instruction, practical skills training will be conducted on mannequins using videolaryngoscopy for intubation. Students who agree to participate will then perform an intubation attempt on a standard airway management mannequin using videolaryngoscopy. Data collected will include demographic characteristics, habits such as video gaming, sports activities, participation in board games like chess, Rubik's Cube, three-dimensional puzzles, and hobbies such as arts and crafts or playing musical instruments. Additionally, parameters such as intubation success (successful/unsuccessful), intubation duration (in seconds), glottic visualization scores (Cormack-Lehane classification and POGO score), and the durations of two specific phases of intubation (glottic visualization time and endotracheal tube passage time) will be recorded.

The study aims to investigate the influence of video game playing habits and certain activities on videolaryngoscopic intubation performance. Glottic visualization will be assessed using the Cormack-Lehane grading system, where Grade I indicates full visualization of the glottis, Grade IIa signifies partial visibility, Grade IIb corresponds to only arytenoid cartilages being visible, Grade III indicates only the epiglottis is seen, and Grade IV denotes no visible glottic structures. The POGO (Percentage of Glottic Opening) score provides a quantitative measure of the proportion of the glottic opening visible during intubation, expressed as a percentage. A POGO score of 100% indicates complete visualization of the glottic opening (from anterior commissure to posterior arytenoids), while a score of 0% indicates no glottic structures are visible (only the epiglottis can be seen). A score of 50% reflects that half of the glottic opening is visible.

The total intubation time is defined as the interval from the beginning of the procedure-placing the laryngoscope blade into the mouth-to the successful placement and confirmation of the endotracheal tube within the trachea. The glottic visualization time refers to the duration from insertion of the laryngoscope into the mouth until the initial clear view of the glottis is obtained. The endotracheal tube passage time is measured from the moment the glottic structures are visualized until the tube passes through the vocal cords into the trachea.

ELIGIBILITY:
Inclusion Criteria:

* Fourth-year medical students undergoing anesthesiology internship
* Those with no previous experience of endotracheal intubation

Exclusion Criteria:

* Those with previous endotracheal intubation experience
* Those with neuromuscular diseases that impair motor function
* Those who have recently undergone hand surgery
* Those who decline to accept the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The primary outcome of our study is the intubation duration. In a previous study, the mean (standard deviation) of intubation time was reported as 90 (45.5) seconds for individuals who played video games and 127.6 (39.5) seconds for those who did not. Considering a two-sided Type I error of 0.05 (95% confidence level), a sample size of 35 participants per group was determined to be sufficient. To account for potential exclusions and dropouts, we plan to include 50 participants in each group, resulting in a total of 100 participants in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Intubation duration | On the day of the manikin-based training session (Baseline, Day 0)
  Intubation duration refers to the period elapsed from the initiation of the procedure, marked by the insertion of the laryngoscope blade into the mouth, to the successful completion of intubation, which is defined as the passage of the endotracheal tube through the vocal cords and its proper placement and verification.

SECONDARY OUTCOMES:
Glottic visualization score | On the day of the manikin-based training session (Baseline, Day 0)
  Glottic visualization during laryngoscopy is quantitatively assessed using the Percentage of Glottic Opening (POGO) score. The POGO score provides an objective measure of the visualized portion of the glottic opening during tracheal intubation. It is expressed as a percentage ranging from 0% to 100%, where 100% indicates full visualization of the glottis-from the anterior commissure to the interarytenoid notch, and 0% denotes that no part of the glottis is visible, with only the epiglottis being seen. Higher POGO scores reflect better glottic visualization.
Intubation success with videolaryngoscopy | On the day of the manikin-based training session (Baseline, Day 0)
  Participant's success or failure in intubation of the manikin using videolaryngoscopy.
Time to visualize the glottis | On the day of the manikin-based training session (Baseline, Day 0)
  The visualization time of the glottis is the time between the introduction of the laryngoscope blade into the mouth and the moment the glottis is clearly seen for the first time.
The transit time of the endotracheal tube | On the day of the manikin-based training session (Baseline, Day 0)
  The tracheal intubation duration refers to the elapsed time from the moment the glottic structures are visualized until the successful placement of the endotracheal tube through the vocal cords into the trachea.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, ABD Veya Kanada'daysanız Lütfen Seçin..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data used to support the findings of this study can be obtained from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For 5 years after the study is completed
Access Criteria: The data supporting the findings of this study are available from the corresponding author upon reasonable request via email.